CLINICAL TRIAL: NCT02280070
Title: Randomized Phase II Study of SOX vs mFOLFOX6 as Neoadjuvant Chemotherapy in Patients With Resectable Rectal Cancer (KSCC1301).
Brief Title: RP II Study of SOX vs mFOLFOX6 in Patients With Resectable Rectal Cancer (KSCC1301).
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Research Support Center Kyush (Other)
Responsible Party: Principal Investigator, Yoshito Akagi, Professor, Kurume University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSCC1301
Record Dates: First submitted 2014-10-16; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Rectal Cancer
Keywords: resectable rectal cancer; SOX; mFOLFOX6; neoadjuvant
MeSH Terms: conditions — Rectal Neoplasms | interventions — Clinical Laboratory Techniques; Hematologic Tests; Blood Chemical Analysis; Health Records, Personal; Restraint, Physical; Body Height; Karnofsky Performance Status; Biomarkers; CA-19-9 Antigen; Hepatitis C Antibodies; Endoscopy; S 1 (combination); Tegafur; gimeracil; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SOX (S-1 + L-OHP) (Active Comparator): S-1 (80 mg/m2, p.o.) (day1-14）, L-OHP (130 mg/m2)(day 1): repeated every 3 weeks until 4 courses or meet discontinuation criteria.
  Medical history and physical examination, BW and height, performance status, laboratory test, creatinine clearance, biomarker, contrasting CT, adverse event, HBs antigen and HCV antibody, endoscopy, HBs antibody and HBc antibody
  Interventions: Other: Laboratory test; Other: Medical history and physical examination; Other: BW and height; Other: Performance status; Other: Creatinine clearance; Other: Biomarker; Radiation: Contrasting CT; Other: Adverse event; Other: HBs antigen and HCV antibody; Other: Endoscopy; Other: HBs antibody and HBc antibody; Drug: S-1; Drug: L-OHP (130mg/m2)
- mFOLFOX6 (Active Comparator): L-OHP (85 mg/m2) and l-LV (200 mg/m2) by IV infusion drip for 2hr at day 1. 5-FU (400 mg/m2) by bolus IV administration just after the L-OHP and l-LV administration. 5-FU (2,400 mg/m2) by IV continuous infusion for 46 hours using infuser pump afterwards (day 1-2: repeated every 2 weeks until 6 courses or meet discontinuation criteria.
  Medical history and physical examination, BW and height, performance status, laboratory test, creatinine clearance, biomarker, contrasting CT, adverse event, HBs antigen and HCV antibody, endoscopy, HBs antibody and HBc antibody
  Interventions: Other: Laboratory test; Other: Medical history and physical examination; Other: BW and height; Other: Performance status; Other: Creatinine clearance; Other: Biomarker; Radiation: Contrasting CT; Other: Adverse event; Other: HBs antigen and HCV antibody; Other: Endoscopy; Other: HBs antibody and HBc antibody; Drug: L-OHP (85 mg/m2); Drug: l-LV; Drug: 5-FU

INTERVENTIONS:
Other: Laboratory test — Leukocyte, neutrophil (ANC ：stab + seg), hemoglobin, platlet, albumin, total birrilubin, AST, ALT, LDH, Creatinine, Na, K, CRP, fast blood sugar
  Other Names: Hematologic test and blood chemistry
Other: Medical history and physical examination — medical history and physical examination
Other: BW and height — Body weight (kg) and height (cm)
Other: Performance status — ECOG performance status, 0: Fully active, able to carry on all pre-disease performance without restriction, 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, 2: Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours, 3: Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours, 4: Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair, 5: Dead
  Other Names: PS
Other: Creatinine clearance — Creatinine clearance (CCr, mL/min) was estimated by Cockcroft & Gault method using serum creatinine (mg/dL), age and body weight (kg).
  Other Names: CCr
Other: Biomarker — Carcinoembryonic antigen and carbohydrate antigen 19-9
  Other Names: CEA and CA19-9
Radiation: Contrasting CT — Computed tomography
  Other Names: CT
Other: Adverse event — AE was evaluated using Common Terminology Criteria for Adverse Events (CTCAE v4.0).
  Other Names: AE
Other: HBs antigen and HCV antibody — check for exclusion criteria
Other: Endoscopy — Endoscopy for lower digestive tract
Other: HBs antibody and HBc antibody — Check according to hepatitis B guideline
Drug: S-1 — S-1 (80 mg/m2, p.o.) is administered at day 1 -14 of the course and repeated every 3 weeks until 4 courses or meet discontinuation criteria.
  Other Names: Tegafur, gimeracil, potassium oteracil potassium
  Arms: SOX (S-1 + L-OHP)
Drug: L-OHP (130mg/m2) — L-OHP (130mg/m2 intravenously) is administered at day 1 of the course and repeated every 3 weeks until 4 courses or meet discontinuation criteria.
  Other Names: Oxaliplatin
  Arms: SOX (S-1 + L-OHP)
Drug: L-OHP (85 mg/m2) — L-OHP (85mg/m2) is administered by IV infusion drip for 2hr at day 1 of the course and repeated every 2 weeks until 6 courses or meet discontinuation criteria.
  Other Names: Oxaliplatin
  Arms: mFOLFOX6
Drug: l-LV — l-LV (200 mg/m2) is administered by IV infusion drip for 2hr at day 1 of the course and repeated every 2 weeks until 6 courses or meet discontinuation criteria.
  Other Names: l-isomer of leucovorin
  Arms: mFOLFOX6
Drug: 5-FU — 5-FU (400 mg/m2) by bolus IV administration just after the L-OHP and l-LV administration. 5-FU (2,400 mg/m2) by IV continuous infusion for 46 hours using infuser pump afterwards and repeated every 2 weeks until 6 courses or meet discontinuation criteria.
  Other Names: 5-fluorouracil
  Arms: mFOLFOX6

SUMMARY:
To evaluate the efficacy and safety of SOX or mFOLFOX6 as neoadjuvant chemotherapy in patients with resectable rectal cancer, and to identify the more promising regimen.

DETAILED DESCRIPTION:
1. Patient registration procedure

If it is confirmed that the subject meets the inclusion criteria and correspondent none of the exclusion criteria, the subject is registered by using CReS Kyushu registration/allocation system (CK-RAS). The registration with CK-RAS is available for 24hr (URL: https://reg.cres-kyushu.or.jp/qmin/login/) and needs for individual ID and password.

2. Quality management

1. Monitoring

   A central monitoring or in-site monitoring are carried out based on the data from case report form (CRF) collecting at data coordinating center. In principle, an on-site monitoring is not carried out, but it may be carried out when the on-site monitoring is determined to need by Kyushu Study group of Clinical Cancer (KSCC) steering committee from the results of the central monitoring so on.
2. Data Monitoring Committee

   A Data Monitoring Committee (DMC) has been established.
3. Data entry

   All data will be entered by the double entry method. Referential data rules, valid values, range checks, and consistency checks against data already stored in the database will be supported. Checks will be applied at the time of data entry into a specific field. Additional errors will be detected by programs designed to detect missing data or specific errors in the data. The investigator who receives the inquiry will respond by checking the original forms for inconsistency, checking other sources to determine the correction, modifying the original paper form entering a response to the query.
4. Regular monitoring report

   A regular monitoring report generated by data coordinating center is submitted to KSCC Steering Committee, principal investigator, the DMC etc and it is reviewed according to "KSCC regulation on the monitoring". The information on the status of site EC approval and the achievement of enrollment: number of enrollment- total/per periodical, total/per site, is reported monthly using e-mail.
   * Contents of monitoring report

     1. Study abstract: schema/purpose/subject/endpoint/definition of treatment/anticipated enrollment number/progress of the study
     2. Enrollment status: per participating site/total
     3. Monitoring activity: contents of activity/CRF collection per site/uncollected CRF, inquiry
     4. Review of the eligible treatment case：the case of ineligible possibility/the case determined as ineligible/number of eligible case/the case determined as non-treatment/total number of treatment case
     5. Review of a target population for analysis: the number of cases targeted for efficacy analysis/safety analysis
     6. Patient background
     7. Treatment time-course: summary of on-treatment and discontinuation/summary of reason for discontinuation/list of reason for discontinuation
     8. Protocol violation/deviation
     9. Safety evaluation: serious adverse reaction, event/the case which was notified to the study group among the adverse reactions, events with an ordinary report/general adverse events
     10. Others
5. Audit

A site audit is carried out by the audit members of KSCC Coordinating Center, data coordinating center, medical staff of other site under the approval of the site director according to "KSCC regulation for site audit". The results of the audit are reported to the site director, KSCC Steering Committee, principal investigator etc. (if required, to DMC).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients who are judged to be suitable for receiving this protocol therapy by physician
* Distal border of tumor is located under the peritoneal reflection
* Histologically confirmed rectal adenocarcinoma
* Previously untreated rectal cancer
* Within 28 days before registration, the tumor is considered by the surgeon to be amenable to curative resection [T category: cSS and cSE, cSI, cA, cAI. N category: cN0-2 and cN3(#253 lymph node)]
* Within 28 days before registration, there is no evidence of distant metastasis by contrast-enhanced CT
* >= 20 years old
* PS (ECOG) 0-1
* Be able to take oral drugs
* Required baseline laboratory parameters (within 14 days before registration): WBC >= 3000 ,<12000/mm3, Neu >= 1,500/ mm3, Hb >= 9.0g/dl, Plt >= 100,000/ mm3, T-Bil <= 2.0mg/dl, AST,ALT <= 100U/L, Cre <1.5mg/dl, Ccr >= 60mL/min
* Considered to survive for more than 3 months

Exclusion Criteria:

* History of serious drug hypersensitivity or a history of drug allergy
* Pregnant or lactating woman and man who hope for Partner's pregnant
* Active infection(over 38 degree)
* Serious complication ( ex. interstitial pneumonitis, pulmonary fibrosis, renal failure, liver failure, serious diabetes, serious hypertension)
* Clinically significant abnormal electrocardiogram or heart disease
* Serious diarrhea
* Pleural effusion, peritoneal fluid that needs treatment
* Previous history of serious lung disorder ( ex. interstitial lung disease or fibrosis, serious emphysema )
* Hemorrhagic diathesis, coagulation disorder
* Active double cancer (synchronous double cancer or asynchronous double cancer with disease-free duration of 5 years or less)
* Patients who need flucytosine, phenytoin or warfarin potassium
* Requiring steroid drug
* Patients with contraindication to therapy
* History of allergy to contrast material
* Serious stricture (exclude the patients who are put in stoma)
* Positive for HBs antigen and HCV antibody
* Not appropriate for the study at the physician's assessment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-09; Primary Completion 2018-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
3-years Disease Free Survival rate | 3 years from the enrollment
  The last analysis after the follow-up period is conducted. The disease-free survival ratio that assumed full analysis set (FAS) as a denominator is estimating by Kaplan-Meier method at 3 year, up to 5 years after the last subject enrollment.

SECONDARY OUTCOMES:
Pathological Effect | After operation, up to 5 years after the last subject enrollment.
  The pathological effect of protocol treatment as FAS a denominator is evaluated according to the criteria of Japanese Classification of Colorectal Carcinoma 7th revision
R0 resection rate | At operation, up to 5 years after the last subject enrollment.
  The R0 resection rate is defined as a ratio of case that conducted R0 resection in FAS.
Completion rate of each modality (neoadjuvant chemotherapy, operation and adjuvant chemotherapy) | After completion of protocol treatment, up to 5 years after the last subject enrollment.
  The rate completed 4 courses of neo-adjuvant chemotherapy within protocol treatment is defined as the completion rate of neo-adjuvant therapy in FAS. Among the cases that an resection operation are enforced and that adjuvant chemotherapy is planned after the operation, the rate completed 4 courses of adjuvant chemotherapy within protocol treatment is defined as the completion rate of adjuvant therapy
Overall survival (OS) | Up to 5 years after the last subject enrollment.
  Overall survival is defined as a period from an enrollment date to a death from every cause in FAS.
Disease Free survival (DFS) | The date of recurrence, occurrence of secondary cancer and death, up to 5 years after the last subject enrollment.
  DFS is defined as the period from a registration day to the day of recurrence, the day of diagnosis of secondary cancer and the day of the death of every cause in FAS.
OS in patients with R0 resection | At the date of death, up to 5 years after the last subject enrollment.
  OS in patients with R0 resection is defined as a period from a enrollment day to the date of death from every cause in patients with R0 resection in FAS.
DFS in patients with R0 resection | The date of recurrence, occurrence of secondary cancer and death, up to 5 years after the last subject enrollment.
  DFS in patients with R0 resection is defined as the period from a enrollment day to the day of recurrence, the day of diagnosis of secondary cancer and the day of the death of every cause in patients with R0 resection in FAS.
Transition rate to Operation | At the operation, up to 5 years after the last subject enrollment.
  The transition rate to operation is defined as the rate of case transited to the resection operation in FAS.
local recurrence rate (per operated population) | After the operation, up to 5 years after the last subject enrollment.
  The local recurrence rate is defined as the recurrence rate of operated population.
Safety | Within protocol treatment, up to 5 years after the last subject enrollment.
  The frequency of worst Grade of the adverse event (toxicity) in all courses with the CTCAE v4.0 Japanese translated JCOG version is calculated in each group about the cases for the safety analysis a denominator
Pattern of first recurrence | At the study completion, up to 5 years after the last subject enrollment.
  Pattern of first recurrence is investigated in FAS.

CONTACTS AND LOCATIONS:
Overall Officials: Yasunori Emi, MD, PhD, Study Director — Saiseikai Fukuoka General Hospital
Locations (2):
- Japan (2):
  - Kyushu University Hospital, Fukuoka
  - Kurume University Hospital, Kurume